CLINICAL TRIAL: NCT04522856
Title: Anaesthesiological Routine Care for Thrombectomy in Cerebral Ischaemia
Status: Recruiting | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: ARCTIC-I
Record Dates: First submitted 2020-06-15; First posted 2020-08-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Ischemia
Keywords: Endovascular thrombectomy; acute ischaemic stroke; large-vessel occlusion
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endovascular thrombectomy: there is only one group of the subjects that had stroke and went under thrombectomy procedure and to see how anaesthesiologists support endovascular thrombectomy with regard to anaesthetic technique,choice of substances, haemodynamic management, and ventilation.

SUMMARY:
Endovascular thrombectomy is the standard of care for acute ischaemic stroke due to large-vessel occlusion. Current guidelines for periprocedural anaesthesiological care give gross recommendations on management of stroke patients during recanalization, but lack detailed information.

To determine how anaesthesiologists support endovascular thrombectomy with regard to anaesthetic technique, choice of substances, haemodynamic management, and ventilation. With a multivariate analysis, the investigators will look for the factors of anesthetic management that are independently correlated with a good or bad outcome.

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* Endovascular stroke treatment involving anaesthesia care

Exclusion Criteria:

* In-hospital onset of stroke
* Inclusion in an interventional study concerning the anaesthesia protocol
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of patients undergoing emergency endovascular thrombectomy for treatment of AIS-LVO. The planned minimum sample size is 5,000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome 90 days after the stroke | 90 days
  Neurological outcome is measured using the modified Rankin Scale [0-6], with higher values indicating worse outcome. As a Primary Outcome Measure, the scale will be dichotomized into good (modified Rankin Scale ≤ 2) versus poor (modified Rankin Scale > 2) outcome.

SECONDARY OUTCOMES:
Mortality | 90 days
  Mortality rate 90 days after the stroke. Mortality rate is the percentage of patients that have died within 90 days following their stroke.
Grade of recanalization | sixty minutes
  Recanalization is classified according to the modified Thrombolysis in Cerebral Infarction classification (mTICI) [0 - 3], with higher values indicating better reperfusion.
Duration | 30 Minutes
  Duration [minutes] from patient's arrival in angiography suite to arterial puncture for endovascular thrombectomy.
  Duration [minutes] from patient's arrival in angiography suite to arterial puncture for endovascular thrombectomy.
  Duration [minutes] from arterial puncture to end of endovascular thrombectomy.
Proportion of patients breathing spontaneously | sixty minutes
  Proportion of patients breathing spontaneously after thrombectomy [Time Frame: On transfer from angiography suite after thrombectomy, which typically takes 1 hour]. This is defined as percentage of patients that breathe spontaneously without laryngeal mask, laryngeal tube, or endotracheal tube after thrombectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ranft, Dr., Study Chair — Senior Physician-München, Germany
Locations (1):
- TU München, München, Germany

IPD SHARING:
Plan to Share IPD: No